CLINICAL TRIAL: NCT01631240
Title: National Health and Nutrition Examination Survey (NHANES), Urinary Sodium Calibration Study
Brief Title: NHANES Urinary Sodium Calibration Study
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011-10
Record Dates: First submitted 2012-06-11; First posted 2012-06-29 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Nutrition Assessment
Keywords: Sodium; Potassium; Iodine; Creatinine

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults 18-39 years: Healthy adults aged 18-39 years

SUMMARY:
This proposed calibration study is designed to evaluate the correlation of urinary sodium excretion between NHANES timed urine and 24-hour urine collections.

DETAILED DESCRIPTION:
The study will be conducted with 400 volunteer participants aged 18-39 years old. Participants will be asked to collect urine samples over a 24-hour period. One-third of the participants (n=133) will be asked to collect a second 24-hour urine 4-11 days later. A 24-hour dietary recall interview will be collected after the completion of each 24-hour urine collection. Results from this study will be used to assess how well the sodium excretion estimated from NHANES timed urine correlates with data from 24-hour urine collection. It will provide valuable information on the potential of NHANES timed urine collections to be used to characterize trends in U.S. population sodium intake.

ELIGIBILITY:
Inclusion Criteria:

English speaking

* Aged 18-39 years old
* 50% Black; 50% all other
* 50% male; 50% female
* At least 50 (25 male; 25 female) of the 400 participants likely to have high sodium diet indicated by selected dietary behaviors
* At least 50 (25 male; 25 female) of the 400 participants likely to have low sodium diet indicated by selected dietary behaviors

Exclusion Criteria:

* Pregnant or trying to get pregnant.
* Taking loop diuretics
* Chronic kidney disease
* New hypertension treatment or change in hypertension treatment in the last 2 weeks

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was conducted with 407 adult volunteer participants living in the Washington DC, Maryland areas who met the following criteria:
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Usual sodium intake | one day
  Usual sodium intake based on 24-hour sodium excretions (two measurements for a one-third subset 4-11 days after the first collection) using measurement error models

SECONDARY OUTCOMES:
Usual potassium intake | one day
  Usual potassium intake based on 24-hour potassium excretions (two measurements for a one-third subset) using measurement error models
Creatinine excretion | one day
  Based on 24-hour creatinine excretion
Usual iodine intake | one day
  Usual sodium intake based on 24-hour sodium excretions (two measurements for a one-third subset 4-11 days after the first collection) using measurement error models

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yih Wang, PhD, Principal Investigator — Centers for Disease Control and Prevention; Mary Cogswell, DrPH, Principal Investigator — Centers for Disease Control and Prevention; Catherine Loria, PhD, Principal Investigator — National Institutes of Health (NIH); Christine Swanson, PhD, Principal Investigator — National Institutes of Health (NIH)

IPD SHARING:
Plan to Share IPD: Yes
Data are available through the NCHS Research Data Center

REFERENCES:
- [Result] Wang CY, Carriquiry AL, Chen TC, Loria CM, Pfeiffer CM, Liu K, Sempos CT, Perrine CG, Cogswell ME. Estimating the population distribution of usual 24-hour sodium excretion from timed urine void specimens using a statistical approach accounting for correlated measurement errors. J Nutr. 2015 May;145(5):1017-24. doi: 10.3945/jn.114.206250. Epub 2015 Apr 1. PMID 25833885
- [Result] Mercado CI, Cogswell ME, Valderrama AL, Wang CY, Loria CM, Moshfegh AJ, Rhodes DG, Carriquiry AL. Difference between 24-h diet recall and urine excretion for assessing population sodium and potassium intake in adults aged 18-39 y. Am J Clin Nutr. 2015 Feb;101(2):376-86. doi: 10.3945/ajcn.113.081604. Epub 2014 Dec 17. PMID 25646336
- [Result] Perrine CG, Cogswell ME, Swanson CA, Sullivan KM, Chen TC, Carriquiry AL, Dodd KW, Caldwell KL, Wang CY. Comparison of population iodine estimates from 24-hour urine and timed-spot urine samples. Thyroid. 2014 Apr;24(4):748-57. doi: 10.1089/thy.2013.0404. Epub 2014 Mar 4. PMID 24308769
- [Result] Cogswell ME, Wang CY, Chen TC, Pfeiffer CM, Elliott P, Gillespie CD, Carriquiry AL, Sempos CT, Liu K, Perrine CG, Swanson CA, Caldwell KL, Loria CM. Validity of predictive equations for 24-h urinary sodium excretion in adults aged 18-39 y. Am J Clin Nutr. 2013 Dec;98(6):1502-13. doi: 10.3945/ajcn.113.059436. Epub 2013 Sep 18. PMID 24047921
- [Result] Wang CY, Cogswell ME, Loria CM, Chen TC, Pfeiffer CM, Swanson CA, Caldwell KL, Perrine CG, Carriquiry AL, Liu K, Sempos CT, Gillespie CD, Burt VL. Urinary excretion of sodium, potassium, and chloride, but not iodine, varies by timing of collection in a 24-hour calibration study. J Nutr. 2013 Aug;143(8):1276-82. doi: 10.3945/jn.113.175927. Epub 2013 Jun 12. PMID 23761643
- [Derived] Freedman LS, Wang CY, Commins J, Barrett B, Midthune D, Dodd KW, Carroll RJ, Kipnis V. Can sodium and potassium measured in timed voids be used as reference instruments for validating self-report instruments? Results from a urine calibration study. Am J Clin Nutr. 2024 May;119(5):1321-1328. doi: 10.1016/j.ajcnut.2024.02.013. Epub 2024 Feb 23. PMID 38403166